CLINICAL TRIAL: NCT05494827
Title: The Impact of a Regular Mineral Water With a High Content of Sodium Bicarbonate (Borjomi®) Consumption on Anaerobic Performance
Brief Title: The Impact of a Regular Borjomi® Consumption on an Anaerobic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zaynudin Zaynudinov, MD, PhD (Other)
Collaborators: LLC IDS Borjomi (Unknown)
Responsible Party: Sponsor-Investigator, Zaynudin Zaynudinov, MD, PhD, Chief physician, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Organization: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 03/20
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Bicarbonate mineral water; Anaerobic performance; Acid-base balance
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant
Masking Description: The intervention (drinking water) was masked for participants through the same indistinguishable bottle design, whereas the taste of the water was different. The research team was unmasked as visits for participants from comparable groups assigned for separate days in order to prevent the possible discussion of water taste between groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Borjomi (Experimental): Healthy volunteers (N16, 8 males and 8 females) 30.63±1.04 y.o. with BMI 22.17±0.75 kg/m2 were randomly allocated to Borjomi group. Participants received 30 bottles (500 ml) of natural mineral water Borjomi® for daily 1000 ml (2 bottles) water consumption for 14 days (from visits 1 and 2). Participants drank the first bottle on the visit 1 after the first study Wingate test and the last bottle on the visit 3 before the second study Wingate test
  Interventions: Other: Regular consumption of natural mineral water Borjomi® with high bicarbonate content
- Smart Spring (Active Comparator): Healthy volunteers (N16, 8 males and 8 females) 28.56±1.61 y.o. with BMI 23.14±0.60 kg/m2 were randomly allocated to Smart Spring group. Participants received 30 bottles (500 ml) of processed drinking water Smart Spring® for daily 1000 ml (2 bottles) water consumption for 14 days (from visits 1 and 2). Participants drank the first bottle on the visit 1 after the first study Wingate test and the last bottle on the visit 3 before the second study Wingate test.
  Interventions: Other: Regular consumption of processed drinking water Smart Spring®
- Control group (Placebo Comparator): Healthy volunteers (N16, 8 males and 8 females) 30.69±1.74 y.o. with BMI 22.67±0.51 kg/m2 were randomly allocated to Control group. Participants received 30 bottles (500 ml) of steal drinking water Святой Источник® for daily 1000 ml (2 bottles) water consumption for 14 days (from visits 1 and 2). Participants drank the first bottle on the visit 1 after the first study Wingate test and the last bottle on the visit 3 before the second study Wingate test.
  Interventions: Other: Regular consumption of still drinking water

INTERVENTIONS:
Other: Regular consumption of natural mineral water Borjomi® with high bicarbonate content — Natural mineral water Borjomi® is a transparent mineral water with specific alkaline taste and smell. The chemical composition includes sodium hydrocarbonate (HCO2-) 3995 mg/l (3500-5000 mg/l), chlorides (Cl-) 360 mg/l (250-500 mg/l), and nitrites (NO2-) <0.005 mg/l (up to 1 mg/l). The "Borjomi" water was packaged into standardized unlabeled 500 ml bottles. Participants were prescribed with 2 bottles (1000 ml) of daily consumption for 14 days. In order to maintain their usual water regimen, the participants additionally consumed steal drinking water on demand. The day before testing, participants were asked to abstain from their routine training and other physical activities.
  Other Names: Borjomi
  Arms: Borjomi
Other: Regular consumption of processed drinking water Smart Spring® — Processed drinking water Smart Spring® has no colour and smell with delicate specific taste. The chemical composition includes sodium (Na+) 33.6 mg/l, magnesium (Mg2+) 10.03 mg/l, calcium (Ca2+) 34.57 mg/l, chlorides (Cl-) 69.79 mg/l, sulfates (SO42-) 22.00 mg/l, and hydrocarbonates (HCO2-) 96.48 mg/l. The Smart Spring® water was packaged into standardized unlabeled 500 ml bottles. Participants were prescribed with 2 bottles (1000 ml) of daily consumption for 14 days. In order to maintain their usual water regimen, the participants additionally consumed steal drinking water on demand. The day before testing, participants were asked to abstain from their routine training and other physical activities.
  Other Names: Smart Spring®
  Arms: Smart Spring
Other: Regular consumption of still drinking water — Still drinking water Святой Источник®is a standard steal drinking water, that has no colour, taste, and smell. The Святой Источник® water was packaged into standardized unlabeled 500 ml bottles. Participants were prescribed with 2 bottles (1000 ml) of daily consumption for 14 days. In order to maintain their usual water regimen, the participants additionally consumed steal drinking water on demand. Participants were asked to abstain from mineral water consumption for the entire observation period.
  Other Names: Water
  Arms: Control group

SUMMARY:
The effects of 2 weeks 1000 ml daily mineral water Borjomy® consumption of anaerobic performance and acid-base balance in comparison with purified electrolite smart-water and still drinking water.

DETAILED DESCRIPTION:
Bicarbonate supplementation increases the efficiency of the body's buffer systems and improves anaerobic performance in athletes when taking bicarbonate just before training. In the course of studies, a similar effect was confirmed for professional swimmers at a distance of 200 meters freestyle, cyclists at distances up to 3 km and track and field athletes in steeplechase. However, these studies were conducted on professional male athletes, and it is interesting to compare the effects with non-athletes population.

Borjomi® is a natural bicarbonate sodium mineral water with high taste qualities. The effects of Borjomi® as bicarbonate source on physical performance are another research interest.

The aim of this study was to evaluate the comparative effectiveness of the regular use of bicarbonate-containing mineral water (Borjomi®) on anaerobic performance and acid-base balance during short-term physical activity of high intensity in comparison with purified electrolite smart-water and still drinking water.

ELIGIBILITY:
Inclusion Criteria:

* Normal body weight (BMI ≥18-24.90 kg/m2).
* Regular physical activity - at least 150 minutes of exercise per week in 2 and more trainings.

Exclusion Criteria:

* Peak oxygen consumption less than 50% of the norm (adjusted for sex and age).
* Allergic reactions to latex.
* Smokers or quit-smokers (less than 6 month of withdrawal).
* Any vitamin, sport or food supplementation in 3 month prior to participation.
* Any low-limb trauma in 6 month prior to participation.
* Any chronic diseases on permanent treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of Relative Peak Power (W/kg) | Twice: Baseline (visit 1) and in 2 weeks (visit 2).
  The Dynamic of Relative Peak Power was evaluated by repeated 30-seconds low limb Wingate anaerobic test with 7.5% from body mass workload in accordance with standard Wingate anaerobic test procedure with individual adjustment of angle and height of handlebar, seat height and foot straps. The test was preceded by a 5 min warm-up with a 4.5% from body mass workload. Wingate anaerobic test were performed by each participant on visit 1 (day 3) and visit 2 (day 16). On visit 0 (day 1) the training Wingate anaerobic test with 4.5% from body mass workload was conducted to familiarize the participants with the testing procedure. The day before testing, participants were asked to abstain from their routine training and other physical activities.
Changes of Fatigue Index (%) | Twice: Baseline (visit 1) and in 2 weeks (visit 2).
  The Fatigue Index was evaluated as percentage of power lost by repeated 30-seconds low limb Wingate anaerobic test with 7.5% from body mass workload in accordance with standard Wingate anaerobic test procedure with individual adjustment of angle and height of handlebar, seat height and foot straps. The test was preceded by a 5 min warm-up with a 4.5% from body mass workload. The day before testing, participants were asked to abstain from their routine training and other physical activities.

SECONDARY OUTCOMES:
Changes of Acid-Base Balance | 6 times: visit 1 - baseline, after Wingate test, and in 5 minutes recovery-period; visit 2 - baseline, after Wingate test, and in 5 minutes recovery-period.
  Cubtal veins were catheterized with Peripheral venous catheters on visits 1 (day 3) and 2 (day 16) before Wingate anaerobic test. The venous blood samples were collected three times in rest, after Wingate anaerobic test, and after 5 minutes recovery-period on visits 1 (day 3) and 2 (day 16). After the last sample collection the catheter was removed (at the same day). The blood samples were immediately analyzed for Acid-Base Balance according to standard laboratory procedures.
Changes of Lactate levels | 6 times: visit 1 - baseline, after Wingate test, and in 5 minutes recovery-period; visit 2 - baseline, after Wingate test, and in 5 minutes recovery-period.
  Cubtal veins were catheterized with Peripheral venous catheters on visits 1 (day 3) and 2 (day 16) before Wingate anaerobic test. The venous blood samples were collected three times in rest, after Wingate anaerobic test, and after 5 minutes recovery-period on visits 1 (day 3) and 2 (day 16). After the last sample collection the catheter was removed (at the same day). The blood samples were immediately analyzed for Lactate levels according to standard laboratory procedures.
Changes of Attention stability | 4 times: visit 1 - baseline and after Wingate test; visit 2 - baseline and after Wingate test.
  Attention stability was assessed in rest and after Wingate anaerobic test on visits 1 (day 3) and 2 (day 16). For attention stability assessment the standard 5x5 Schulte Table testing with calculation of work efficiency, work warm-up and psychological stability was used.

CONTACTS AND LOCATIONS:
Overall Officials: Zaynudin M. Zaynudinov, Dr, Principal Investigator — Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Locations (1):
- Department of Cardiovascular Pathology and Diet Therapy of Nutrition Clinic of The Federal Research Centre of Nutrition, Biotechnology and Food Safety, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
The whole data set was shared with LLC IDS Borjomi (funding provider) after personal data (name, 2nd name and surname) were changed to individual participants numbers (ID).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data set was shared at December 2020 after the study completion.
Access Criteria: Anonymous data set was shared for statistical analysis, manuscript preparation and power calculations of future research projects.